CLINICAL TRIAL: NCT04443868
Title: Double-Blinded, Placebo-Controlled Parallel, Phase II Clinical Efficacy Study Evaluating NORS To Treat and Prevent the Exacerbation of Infection in Individuals With Documented Mild COVID-19
Brief Title: Nitric Oxide Releasing Solution to Treat and Prevent Exacerbation of Mild COVID-19 Infection
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No subjects enrolled
Sponsor: Sanotize Research and Development corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: COVID-IND-02
Record Dates: First submitted 2020-06-20; First posted 2020-06-23 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-07

CONDITIONS: SARS-CoV Infection
MeSH Terms: conditions — Severe Acute Respiratory Syndrome | interventions — Nitric Oxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nitric Oxide Releasing Solution (Experimental): Daily nasal irrigation (240mL) 14.4ppm
  Interventions: Drug: Nitric Oxide-Releasing Drug
- Placebo Isotonic Saline (Placebo Comparator): Daily nasal irrigation (240mL) 0.9% saline
  Interventions: Drug: Nitric Oxide-Releasing Drug

INTERVENTIONS:
Drug: Nitric Oxide-Releasing Drug — Nasal Spray + Nasal Irrigation
  Other Names: nitric oxide

SUMMARY:
This is a double-blinded, placebo-controlled parallel, phase II clinical efficacy study evaluating Nitric Oxide Nasal Irrigation (NONI) for the treatment of COVID-19 in individuals with mild COVID-19 Infection.

DETAILED DESCRIPTION:
Up to 50 subjects will be enrolled into one of two cohorts of this study in a ratio of 1:1 (Treatment: Placebo Control). Subjects will be screened and randomized into one of two parallel cohorts.

* Treatment (N = up to 25): Subjects will be enrolled and receive daily NONI treatment for 14 days with a follow-up visit on Day 28 post randomization.
* Placebo (N = up to 25): Subjects will be enrolled and receive a placebo for 14 days with a follow-up visit on Day 28 post randomization.

ELIGIBILITY:
Inclusion Criteria:

* Capable of understanding and providing signed informed consent and ability to adhere to the requirements and restrictions of this protocol;
* Men and Women ≥ 18years of age;
* Internet access and capability and willingness to use to participate in audio or audio/video engagements with medical professionals, receive texts, emails, and phone calls from study staff and have a device and reasonable cellular data or other internet access to submit daily study required information using a smart phone, tablet, laptop, or desktop computer during the study period;
* COVID-19 infection confirmed with a laboratory antigen or SARS-CoV-2 RT-PCR nasal swab;
* Specimen collected within the past 48 hours;
* Mild COVID /FLU symptoms which may include no symptoms, fever, cough, sore throat, malaise, headache, muscle pain, gastrointestinal symptoms, lack of taste or smell without shortness of breath or dyspnea;
* Must be willing to use one highly effective birth control method which include: abstinence, hormonal contraceptives (e.g. combined oral contraceptives, patch, vaginal ring, injectables, and implants); intrauterine device (IUD) or intrauterine system (IUS); vasectomy and tubal ligation or to use two forms of effective birth control methods which include: barrier methods of contraception (e.g. male condom, female condom, cervical cap, diaphragm, contraceptive sponge);

  * Hormonal methods and the IUD must be in use at least 30 days prior to first Study drug administration
  * Abstinence and barrier methods must be in use at least 14 days prior to Study drug administration
  * Vasectomy must be completed 3 months prior to first Study drug administration; or in the alternative that a 0 sperm count will suffice.

Exclusion Criteria:

* Current tracheostomy or laryngectomy;
* Concomitant respiratory therapy such as oxygen or ventilatory support. Positive airway pressure for obstructive sleep apnea is permitted if treatment was established with good compliance at least 3 months before enrolment;
* Need for hospitalization for any reason;
* Inability to safely self-administer nasal irrigation
* Any clinical contraindications, as judged by the Qualified Medical Practitioner;
* Clinical signs indicative of moderate, severe or critical COVID severity symptoms (as defined by FDA COVID-19 Guidance Document)
* Mentally or neurologically disabled patients who are considered not fit to consent to their participation in the study;
* Lactating, pregnant or planning to become pregnant during the study period;
* Diagnosed with prior COVID-19 infection (>48 hours from the time the test is reported prior to the time of screening).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
To Measure the efficacy of NONI compared to saline placebo control to shorten the duration of COVID-19 viral infectivity | 6 Days
  Measure the SARS-CoV-2 viral load (Cycle threshold) at baseline through Day 6 between NONI and control arms.

SECONDARY OUTCOMES:
To Measure the virucidal effect of NONI compared to placebo in the nasal cavity in subjects with mild COVID-19 infection | 2, 4 and 6 days
  Measure the proportion of subjects reaching Ct threshold (ie: unmeasurable viral load) between NONI and control
To Measure the virucidal effect of NONI compared to placebo in the nasal cavity in subjects with mild COVID-19 infection | 2, 4 and 6 days
  Measure the difference in time-to Ct threshold (ie: unmeasurable viral load) between NONI and control.
To Measure the efficacy of NONI in prevention of progression of COVID-19 | 28 days
  Measure the proportion of subjects requiring hospitalization or ER/ED visits for COVID-19/flu-like symptoms
To measure reduction of patient reported outcome (PRO) of clinical cold score symptoms and quality of life (QoL) in subjects with COVID-19 | 6 days
  Measure the difference in 12-point COVID Symptom PROs score 0-3 (min 0 & max 36) and a QoL score from 0-100 (lower is worse) from baseline between NONI and control arms.
To measure reduction of patient reported outcome (PRO) of clinical cold score symptoms and quality of life in subjects with COVID-19 | 2, 4, 6, 14 and 28 days
  Measure the difference in proportion of subjects experiencing a reduction of ≥ 5 from baseline between NONI and control arms.
To measure reduction of patient reported outcome (PRO) of clinical cold score symptoms and quality of life in subjects with COVID-19 | 2, 4, 6, 14 and 28 days
  Measure the difference in proportion of subjects with reduction to a score of zero from baseline between NONI and control arms.
To measure the tolerance of NONI compared to saline placebo in participants with mild COVID-19 infection | 14 days
  Number of participants lost-to-follow-up,discontinuing study treatment or number of treatments due to intolerance
To measure the tolerance of NONI compared to saline placebo in participants with mild COVID-19 infection | 14 days
  Severity and frequency of adverse events, pain, discomfort or discontinuations of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Mike armstrong, MD, Principal Investigator — Richmond ENT; Chris Miller, Ph.D, Study Director — SaNOtize Scientific Advisor

IPD SHARING:
Plan to Share IPD: No